CLINICAL TRIAL: NCT07381595
Title: Impact of Subgingival Instrumentation on Clinical and Immunohistochemical Presentation of Oral Lichen Planus With Gingival Involvement
Brief Title: Role of Subgingival Instrumentation in Oral Lichen Planus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRU2025807
Record Dates: First submitted 2025-12-04; First posted 2026-02-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Oral Lichen Planus
Keywords: Subgingival instrumentation; Immunohistochemistry; CD4 and CD8 lymphocytes; Clinical parameters
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Lichen Planus (Experimental): Scaling and root planing will be conducted on Oral Lichen Planus cases with gingival involvement.
  Interventions: Procedure: subgingival instrumentation

INTERVENTIONS:
Procedure: subgingival instrumentation — Subgingival instrumentation like scaling and root planing of the recruited subject shall be done.

SUMMARY:
The goal of this interventional study is to assess the clinical and histopathological changes in Oral Lichen Planus patients with gingival involvement pre and post subgingival instrumentation.

Objective- Primary objective: To observe and evaluate the clinical signs and symptoms in Oral Lichen Planus with gingival involvement. Secondary objective: To observe and evaluate the Cluster of Differentiation (CD) 4+ and 8+T lymphocytes in Oral Lichen Planus with gingival involvement.

Study group: 30 cases of Oral Lichen Planus with gingival involvement

DETAILED DESCRIPTION:
Title: Impact of subgingival instrumentation on clinical and immunohistochemical presentation of Oral Lichen Planus with gingival involvement.

It aims to answer whether subgingival instrumentation will lead to a reduction in clinical signs and symptoms, as well as a decrease in the immunohistochemical expression of Cluster of Differentiation (CD) 4+ and CD8+T lymphocytes. P-(Population)- Oral Lichen Planus patients with gingival involvement. I (Intervention)- Root planing and scaling. C (Comparison)- Same cases after 4 weeks. O (Outcome)- Assessment of clinical symptoms, pain and gingival index at baseline and after 4 weeks. Quantitative assessment of CD4+ and CD8+T lymphocytes at baseline and after 4 weeks.

Periodontitis is an irreversible plaque-induced microbial disease that leads to the destruction of the periodontal ligament and alveolar bone. Its etiopathogenesis is multifactorial and controversial. Oral lichen planus is a T-cell mediated chronic mucocutaneous disease of unknown etiology with an impact of 0.1-4% of the general adult population. Despite various pharmacological advances, the medical management of oral lichen planus remains a daunting task. This could be attributed to the fact that the etiopathogenesis of this disease remains unascertained. Recent evidence does show interactions between these two diseases, where some researchers found that periodontal status in oral lichen planus cases was significantly worse than in healthy controls. Other reports stated that in gingival atrophic-erosive-type oral lichen planus lesions, there was a significant increase in dental plaque and calculus deposits, associated with a higher incidence of periodontal deterioration. Cumulative evidence supports the role of immune dysregulation mediated by the release of cytokines by activated T cells. There is evidence that effective plaque control diminishes the gingival lesions of oral lichen planus, which could be improved by the maintenance of proper oral hygiene and periodontal treatment. However, whether this change in symptoms also makes any histological difference is yet to be known.

To date, no study has evaluated the role of T lymphocytes (CD 8+ cytotoxic & 4+ helper) pre and post scaling and root planing in cases of oral lichen planus with gingival involvement. This study was conceived to evaluate the change in clinical signs and symptoms in oral lichen planus with gingival involvement, as well as a reduction in the number of CD4+ and CD8+T lymphocytes pre and post-treatment.

ELIGIBILITY:
Inclusion criteria:

* Clinically and histopathologically confirmed cases of OLP.
* OLP predominantly involving the gingiva.
* Consent obtained.

Exclusion criteria:

* Cases which does not fulfil either clinical or histopathological criteria.
* Unwilling to participate in the study.
* Patients with recorded history of factors that might modify immune response (such as patient on corticosteroids or medically compromised patients or suffering from heart diseases).
* Cases undergoing treatment of OLP within past 6 months.
* Biopsies with inadequate or non-representative samples
* Cases histopathologically diagnosed as Lichenoid Dysplasia or Oral Lichenoid Lesions.
* Cases diagnosed with autoimmune disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinical signs and symptoms in cases of oral lichen planus | At baseline and after end of treatment at 4 weeks
  Clinical signs and symptoms will be recorded using oral disease severity score criteria

SECONDARY OUTCOMES:
Change in the number of CD4+ and CD8+T lymphocyte count pre and post-treatment in cases of oral lichen planus | At baseline and after end of treatment at 4 weeks
  Each case will be biopsied, the tissue will be processed and quantified for CD4 and CD8 lymphocytes by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India